CLINICAL TRIAL: NCT07124156
Title: A Randomised Phase Ib Trial to Assess the Blood-stage Efficacy of SUM-101 Malaria Vaccine in Adults Residing in Malaria-endemic Settings, After Controlled Human Malaria Infection Using 3D7 P. Falciparum Blood-stage Malaria Infection
Brief Title: A Challenge Study to Assess the Blood-stage Efficacy of Full-length SUM-101 Malaria Vaccine Candidate
Acronym: CHMI-SUM-101
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: European Vaccine Initiative (Other)
Collaborators: Luxembourg Institute of Health (Other Government); Ifakara Health Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVI-CT-002
Record Dates: First submitted 2025-07-04; First posted 2025-08-15 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-07

CONDITIONS: Malaria Fever
Keywords: SUM-01; CHMI; Malaria
MeSH Terms: conditions — Malaria | interventions — 1-acetyl-1,2,3,3a,8,8a-hexahydro-8a-hydroxy-5-methoxypyrrolo(2,3-b)indole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three dose SUM-101 (Experimental): Twelve participants will receive three monthly inoculations (on D0, D28 and D56) with the IMP, SUM-101.
  Interventions: Biological: SUM-101; Other: CHMI
- Three dose Verorab (Active Comparator): 12 participants will receive three monthly inoculations (on D0, D28 and D56) with the IMP Verorab®
  Interventions: Other: CHMI; Biological: Verorab®

INTERVENTIONS:
Biological: SUM-101 — Once randomised to either the SUM-101 or the rabies control vaccine, the participant will always receive the same dose of the same compound (150 µg MSP1 protein dissolved in 0.9% NaCl with 250 µl (5µg) of adjuvant GLA-SE and there are no dose adjustments foreseen. The three vaccine doses will be applied in 4-week intervals on day 0, day 28 and day 56.
  Arms: Three dose SUM-101
Other: CHMI — Experimental intervention: The participants will receive a target dose of 2,800 viable intraerythrocytic P. falciparum 3D7 parasites, in a volume of 2 mL injectable saline. The erythrocytes will be thawed, resuspended and viability will be calculated. The total erythrocyte number will be between ~3.9×106 and ~5.2×108 (average: ~4.55×108) per dose with ≥80% (~3.64×108) P. falciparum ring-stage parasites and around 34% (~1.24×108) viability. This number of viable P. falciparum ring-stage parasites will be diluted to establish 2800 per syringe that will be administered. Challenge dose will be administered to all volunteers as an intravenous injection at the clinical site following instructions in an established SOP. The parasites injected in each volunteer will be quantified retrospectively using qPCR analysis.
  The parasites injected in each volunteer will be quantified retrospectively using qPCR analysis. No dose adjustments are foreseen. As described in the protocol
Biological: Verorab® — Once randomised the participant will receive the or Verorab® and there are no dose adjustments foreseen. The three vaccine doses will be applied in 4-week intervals on day 0, day 28 and day 56.
  Arms: Three dose Verorab

SUMMARY:
The goal of the study is to test the efficacy using a homologous CHMI of this vaccine candidate early in the development path in a population living in malaria-endemic areas.

In the previous Phase Ia and Ib trials, no efficacy endpoints were defined, and therefore there is currently no data on the SUM-101 vaccine efficacy. The proposed clinical trial will enrol malaria pre-exposed healthy adults and will be the second trial where the IMP will be administered to healthy adult participants in Tanzania with some pre-existing immunity against malaria.

The vaccination part of this study will be performed in a randomised, double-blinded, controlled design to evaluate the safety, reactogenicity and immunogenicity of the candidate malaria vaccine SUM-101 (MSP1 with GLA-SE as adjuvant). Given that SUM-101 is a malaria vaccine with an important blood-stage component, we propose to use CHMI with the 3D7 P. falciparum strain-infected red blood cells to establish initial vaccine efficacy data after the third vaccination in a malaria-exposed population.

DETAILED DESCRIPTION:
Full-length MSP1/GLA-SE (SUM-101) malaria vaccine (formerly SumayaVac-1) has been developed by Sumaya Biotech, a spin-off from Heidelberg University, Germany. SUM-101 is a vaccine based on the 3D7 strain (D-form) of full-length merozoite surface protein 1 (full-length MSP1). The full-length MSP1 is expressed as a recombinant heterodimeric protein in E. coli and lyophilised at 150 μg/vial. The lyophilised MSP1 protein is stored at 2 - 8°C. The adjuvant, GLA-SE, was developed by Access to Advanced Health Institute (AAHI), a Washington non-profit corporation with offices at 1616 Eastlake Ave. E, Suite 400, Seattle, WA 98102, USA. It is a stable oil-in-water emulsion containing a synthetic analogue of bacterial glucopyranosyl lipid A and functions as a toll-like receptor 4 agonist. A vial of the adjuvant contains 20μg of GLA-SE in a 400μl emulsion. GLA-SE adjuvant and emulsion formulations should be stored at 2 - 8°C.

The vaccine (SUM-101) is prepared before administration by reconstituting the lyophilised protein in saline (aqueous 0.9% NaCl) and then combining it with the GLA-SE adjuvant. The formulated vaccine is stable at room temperature for up to 60 minutes and administered intramuscularly.

A Phase I first-in-human, double-blinded, randomised trial (PMC6994672) was conducted to assess the safety and immunogenicity of SUM-101 in healthy malaria-naïve adult volunteers in Heidelberg, Germany. The trial demonstrated that SUM-101 is safe, with no serious adverse events (SAE) reported. Vaccination with SUM-101 induced MSP1 specific IgG and IgM antibodies that activated Fc-mediated effector mechanisms and were equally reactive against the vaccine variant (MSP1D/3D7) and a heterologous variant of MSP1 (MSP1F/FCB1). In addition, a Phase Ib trial was conducted in Bagamoyo, Tanzania (NCT05644067, data not yet published) where 20 healthy Tanzanian adults were vaccinated with SUM-101. Preliminary results indicate that SUM-101 is safe and well-tolerated in healthy African adults living in malaria-endemic areas, with ongoing assessments of antibody responses.

Concurrently with this trial, a Phase Ib, randomised, controlled age de-escalation, dose-finding study to evaluate the safety, reactogenicity and immunogenicity of full-length MSP1/GLA-SE (SUM-101) malaria vaccine in healthy young children, and infants (NCT06618885) will be conducted in Burkina Faso. The protocol has been submitted for ethical and regulatory approval in Burkina Faso.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any study procedure.
* Literate participants aged ≥18 - ≤45 years of African origin.
* Female and male participants willing to practice effective contraception from 4 weeks before 1st vaccination (female participants only) and up to 12 weeks after the last vaccination or CHMI (female and male participants)
* Female participants must be willing to undergo multiple serum pregnancy tests.
* Available to participate in follow-up for the duration of the study, including the CHMI in-patient confinement period.
* Contactable by phone during the whole study period.
* At least two years of residence in the Bagamoyo district or nearby districts in the Coastal and Dar-es-Salaam regions and planning to reside there for at least 9 more months.
* Agreement to provide personal contact information and contact information of another household member or close friend.
* Confirmation of understanding of design, procedures, risks and benefits of the study by scoring 10 out of 10 in a structured ten questions with a maximum of two attempts.
* General good health based on assessment of medical history and clinical examination.
* The volunteer agrees to refrain from blood donation for 12 months following CHMI.
* Volunteer agrees to refrain from intensive physical exercise (disproportionate to the volunteer's usual daily activity or exercise routine) during the malaria challenge period.

Exclusion Criteria:

* Previous participation in any malaria vaccine trial in the last 3 years.
* Participation in any other clinical trial involving investigational medicinal products within 30 days prior to the screening assessment.
* Previous history of drug or alcohol abuse interfering with normal social function within one year prior to enrolment.
* Previous vaccination with a rabies vaccine.
* High anti-schizont antibody level as measured by ELISA at screening.
* Intake of chronic medication, especially immunosuppressive agents (steroids, immunomodulating drugs) during the 13 weeks preceding the screening visit or during the study period.
* Known hypersensitivity to any of the vaccine components (adjuvant or protein) or anti-malarial treatments.
* Body mass index (BMI) of ≤18 or ≥30 Kg/m2.
* Participants are unable to be closely followed for social, geographic or psychological reasons.
* Any vaccination from 4 weeks prior to the 1st vaccination and (none planned) up to 8 weeks after the 3rd vaccination.
* Any history, or evidence at screening, of clinically significant symptoms, physical signs or laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, neurological, psychiatric, allergy, endocrine, malignant, haematological, infectious disease, epilepsy and other conditions, which could interfere with the interpretation of the trial results or compromise the health of the participants.
* Abnormal electrocardiogram on screening: pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, clinically significant arrhythmias, left bundle branch block, secondary or tertiary A-V (atrio-ventricular) heart block.
* Any clinically significant laboratory values at screening outside of normal ranges for study participants.
* Malaria positivity at screening (microscopy or qPCR positive).
* Positive HIV, Hepatitis B (HBV) or Hepatitis C (HCV) tests. (The testing will only be requested on the discretion of clinician)
* For females: Positive pregnancy test or actively breastfeeding.
* Any recent or current systemic therapy with an antibiotic or drug with potential antimalarial activity (chloroquine, doxycycline, tetracycline, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, erythromycin, hydroxychloroquine, etc.) (allowable time frame for use at investigators discretion or within a month prior to 1st vaccination or CHMI )
* History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
* Known hypersensitivity to or contra-indications (including co-medication) for use of chloroquine, artemether-lumefantrine, Primaquine or history of severe (allergic) reactions to blood transfusion.
* Being an employee or relative of an employee of Ifakara Health Institute.
* Any other condition or situation that would, in the opinion of the investigator, place the volunteer at an unacceptable risk of injury or render the volunteer unable to meet the requirements of the protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy- Time to diagnosis | From Day 84 to Day 168
  Blood-stage efficacy of the SUM-101 vaccine against 3D7 clone parasites in a CHMI model in healthy malaria-exposed adult volunteers, measured as time to diagnosis in the vaccine arm compared to controls. Time to diagnosis is defined as the number of days from challenge to treatment
Frequency of local and systemic solicited adverse events | After each vaccination (done on Day 0, Day 28 and Day 56) up to 7 days post-vaccination
  Safety of SUM-101 vaccine in healthy malaria-exposed adults as assessed by the frequency of local and systemic solicited adverse events (AEs)
Frequency of local and systemic unsolicited adverse events | After each vaccination (done on Day 0, Day 28 and Day 56) up to 28 days post-vaccination
  Safety of SUM-101 vaccine in healthy malaria-exposed adults as assessed by the frequency of local and systemic unsolicited adverse events
Frequency of any serious adverse events (SAE) | Baseline (Day 0 before 1st vaccination) to end of the follow up (Day 168)
  Safety of SUM-101 vaccine in healthy malaria-exposed adults as assessed by any serious adverse events (SAE)
Number of participants with treatment-related adverse events as assessed by safety laboratory measures of haematology and biochemistry. | Baseline (Day 0 before 1st vaccination) to end of the follow up (Day 168)
  Number of participants with treatment-related adverse events as assessed by safety laboratory measures of haematology and biochemistry.
  Changes in laboratory safety parameters as summarised as absolute values of:
  Haematology: Haemoglobin, WBC (differentiation of eosinophils and neutrophils), platelets and haematocrit.
  Biochemistry: parameters at screening will include: ALT, AST, total bilirubin, creatinine and glucose (random). Troponin sample will be collected before 1st vaccination (at baseline) and stored to be run retrospectively if needed in case of a cardiac event. The sample collected at the time of the cardiac event will be compared with the sample collected at baseline.
  Urinalysis performed by dipstick. Proteinuria, glucose and blood.
MSP1-specific IgG antibody levels assessed by ELISA | Day 0 (pre-vaccination) and Day 84 (Pre-CHMI).
  Humoral immunogenicity of SUM-101 in malaria-exposed adults assessed as MSP1-specific IgG antibody levels measured by serum ELISA in sera collected at Day 0 (pre-vaccination) and Day 84 (Pre-CHMI).

SECONDARY OUTCOMES:
Immunogenicity to MSP1-specific IgM antibody levels measured by ELISA | Day 0 (pre-vaccination) and Day 84 (Pre-CHMI).
  Humoral immunogenicity of SUM-101 in malaria-exposed adults assessed as MSP1-specific IgM antibody levels measured by serum ELISA in sera collected at Day 0 (pre-vaccination) and Day 84 (Pre-CHMI).
Immunogenicity assessed as antibody-mediated complement fixation activity. | Day 0 (pre-vaccination) and Day 84 (Pre-CHMI)
  Humoral immunogenicity of SUM-101 in malaria-exposed adults assessed as antibody-mediated complement fixation activity.
Antibody-mediated complement fixation activity | Day 0 (pre-vaccination) and Day 84 (Pre-CHMI)
  Humoral immunogenicity of SUM-101 in malaria-exposed adults assessed as antibody-mediated complement fixation activity.
Antibody-dependent respiratory burst (ADRB) activity | Day 0 (pre-vaccination) and Day 84 (Pre-CHMI)
  Humoral immunogenicity of SUM-101 in malaria-exposed adults assessed as antibody-dependent respiratory burst (ADRB) activity.

OTHER OUTCOMES:
Comparison of P. falciparum in vivo parasite growth rates | Day 84 to Day 168
  Blood-stage efficacy of SUM-101 malaria vaccine candidate against 3D7 clone parasites in a CHMI model in healthy malaria-exposed adult volunteers, assessed as a comparison of P. falciparum in vivo parasite growth rates (such as parasite multiplication rate, maximum parasitemia, area under the curve, HRP2 levels or total parasites calculation and other outcomes based on parasite growth) in SUM-101 versus Verorab® arm.

CONTACTS AND LOCATIONS:
Overall Officials: Ally Olotu, MD, Principal Investigator — Ifakara Health Institute (IHI)

IPD SHARING:
Plan to Share IPD: No